CLINICAL TRIAL: NCT04789343
Title: The Effect of Reciprocating Instrument and Obturation Techniques on Postoperative Pain in Retreatment : A Prospective Clinical Study
Brief Title: The Effect of Instrumentation and Obturation on Postoperative Pain in Retreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAG-C-DUP-170419-0144
Record Dates: First submitted 2021-02-23; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Endodontically Treated Teeth; Post Operative Pain
Keywords: post operative pain, retreatment
MeSH Terms: conditions — Tooth, Nonvital; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Conventional root canal treatment was perfomed to 45 patients who had been done unacceptable root canal treatment (such as short root canal filling ) on lower premolar or molar teeth before. The patents were healthy and did not take any antibiotics or any medication .
Who Masked: Participant
Masking Description: The patients asked one of three numbers (1-2-3) before treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- hand files with lateral condensation technique (Experimental): Previously done root canal filling removed by hand files (Hedstrom file,VDW, Munich,Germany ) and shaped with the same files and after instrumentation, all canals were filled by AH Plus sealer (Dentsply De Tray, Costanz, Germany) and lateral condensation technique of gutta-percha.
  Interventions: Other: Root canal treatment
- Reciproc instrument with lateral condensation technique (Experimental): Previous root canal filling removed by Reciproc instrument (VDW ,Munich, Germany )using Endomotor (VDW, Munich, Germany). After removal, root canal instrumented with the same instrument and obturated using AHPlus sealer with lateral condensation technique of gutta-percha.
  Interventions: Other: Root canal treatment
- Reciporoc instrument with continuous warmed condensation technique (Experimental): Previous root canal removed by Reciproc instrument using Endomotor, shaped and obturated by AhPlus sealer with continuous gutta-percha technique (Diadent Dia-Duo (Diadent, Chongju, Korea).
  Interventions: Other: Root canal treatment

INTERVENTIONS:
Other: Root canal treatment — The patient usually takes anaesthesia before treatment and access cavity was prepared on the tooth and root canal removed and instrumented and obturated. However, in the present study, previously done root canal was retreated. Usually no anaesthesia was used because all root canals were done before. So just instrumentation and obturation was done.

SUMMARY:
Objectives: The aim of this study was to assess postoperative pain in prospective randomized clinical trial comparing Reciproc or hand instrument and also different obturation techniques in one visit of endodontic retreatment.

Conventional root canal treatment was done to 45 patients who needed retreatment. All instruments used in this study are routinely used instrument in endodontic therapy. After completed root canal treatment, the patients asked the intense of post operative pain.

DETAILED DESCRIPTION:
Materials and metods: The study was included 45 patients (18-65 yrs old) who needed endodontic retreatment in mandibular premolar or molar without any symptoms. The teeth had been randomly assign into 3 groups according to the instrumentation or obturation techniques; hand files with lateral condensation, Reciproc with lateral condensation, or Reciproc with continuous condensation technique. Retreatments had performed in a single visit. Coronal restorations were removed, the gutta-percha were extracted using either Reciproc or hand files. After, biochemical and mechanical praparation, the canals were filled with gutta-percha cones and AH Plus sealer using the lateral condensation or continuous wave of obturation technique. Participants were been asked to rate the incidence and intensity of the postoperative pain on a verbal rating scale 24h, 48h and 72h and 7 days after retreatment. All data were analyzed using (Chi-square test, p=0,05)

ELIGIBILITY:
Inclusion Criteria:

* patients who had previosly done unacceptable root canal treatment on lower premolar or molar with no pain.

No medication should be taken 10 days before treatment for any reason ( such as corticosteroid, antibiotics or analgesic )

Exclusion Criteria:

* age less than 18 or over 65,pregnancy nonrestorable tooth other than lower molar or premolar tooth with more than 4mm periodontal pocket root with broken instrument or any post

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-29 (Actual)

PRIMARY OUTCOMES:
Post operative pain | 24 hours.
  VRS scale was used to assess the intensity of post operative pain or discomfort( 0: no pain,1:mild pain, no medication (analgegic) is requiered, 2 :moderate pain ,feeling pain but no medication is required, 3: severe pain: feeling pain need to take analgesic

SECONDARY OUTCOMES:
Post operative pain; change is being assessed. | 48 hours
  VRS scale was used to assess the intensity of post operative pain or discomfort( 0: no pain,1:mild pain, no medication (analgegic) is requiered, 2 :moderate pain ,feeling pain but no medication is required, 3: severe pain: feeling pain need to take analgesic

OTHER OUTCOMES:
Post operative pain; change is being assessed. | 72 hours.
  VRS scale was used to assess the intensity of post operative pain or discomfort( 0: no pain,1:mild pain, no medication (analgegic) is requiered, 2 :moderate pain ,feeling pain but no medication is required, 3: severe pain: feeling pain need to take analgesic
post operative pain; change is being assessed. | 7 days.
  VRS scale was used to assess the intensity of post operative pain or discomfort( 0: no pain,1:mild pain, no medication (analgegic) is requiered, 2 :moderate pain ,feeling pain but no medication is required, 3: severe pain: feeling pain need to take analgesic

CONTACTS AND LOCATIONS:
Overall Officials: Hesna Sazak Ovecoglu, DDS, PhD, Study Chair — Marmara University Faculty of Dentistry Department of Endodontics
Locations (1):
- Marmara University Faculty of Dentistry, Basibuyuk Campus, Maltepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All statistical datas was documented in post doctorate thesis and will be available at www.tez.gov.tr in a month. Also will be send for publication in one of the dental journal.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Approximately 1 month later in www.tez.gov.tr
Access Criteria: by the title of the study or the name of the researchers